CLINICAL TRIAL: NCT01170936
Title: An Open-label Pilot Study to Assess the Efficacy and Safety of a Single Dose Regime of Canakinumab (ACZ885) in Patients With Active, Refractory Urticarial Vasculitis
Brief Title: Ilaris® in Urticarial Vasculitis - Investigation of Treatment Responses
Acronym: ILUVIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Karoline Krause, Karoline Krause, MD, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILUVIT1; 2010-020063-21 (EudraCT Number)
Record Dates: First submitted 2010-07-26; First posted 2010-07-28 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Urticaria; Vasculitis
Keywords: Urticarial vasculitis; anti-IL1ß therapy
MeSH Terms: conditions — Urticaria; Vasculitis | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Canakinumab (Experimental)
  Interventions: Drug: canakinumab

INTERVENTIONS:
Drug: canakinumab — Single dose of canakinumab 300mg s.c. injection
  Other Names: Ilaris

SUMMARY:
This is a single-center open label study to assess the efficacy and safety of single doses of canakinumab (trade name Ilaris®), a high-affinity monoclonal antibody that neutralizes IL-1β, in patients with active urticarial vasculitis. Efficacy is primarily assessed by a combined symptom score, the urticarial vasculitis activity score (UVAS). Following a baseline period of 2 weeks, patients will be dosed with two single s.c. injections of 150 mg (consistent with a total dose of 300 mg canakinumab). Visits for investigator's assessments will be scheduled at 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks and 16 weeks post dose. Patient's self-assessment will be performed on a daily basis throughout the study. Overall a max. of 10 subjects with urticarial vasculitis will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* UV diagnosis based on diagnostic criteria defined in Appendix 3
* Active UV, refractory to treatment with antihistamines, NSAIDS or colchicine, hydroxychloroquine or dapsone
* Patients who have a mean symptom score (UVAS) of at least 5 during baseline
* If necessary, concurrent/ongoing treatment with a stable dose of systemic corticosteroids not greater than 10mg/d for 14 days prior to screening
* If necessary, concurrent/ongoing treatment with a stable dose of antihistamines and NSAIDs for 7 days prior to screening
* Informed consent signed and dated
* Able to read, understand and willing to sign the informed consent form and abide with study procedures
* Willing, committed and able to return for all clinic visits and complete all study-related procedures, including willingness to have SC injections administered by a qualified person
* In females of childbearing potential: Negative pregnancy test; males and females willing to use highly effective contraception (Pearl-Index < 1). A woman will be considered not of childbearing potential if she is post-menopausal for greater than two years or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy)
* In men: Willingness to utilize highly effective contraception and to not have their partner become pregnant during the full course of the study. Adequate contraceptive measures include oral contraceptives (stable use for two or more cycles prior to screening); bilateral tubal ligation; vasectomy; condom or diaphragm plus either contraceptive sponge, foam or jelly
* Subjects are considered eligible, if they meet the following tuberculosis (TB) screening criteria: no history of latent or active TB prior to screening, no signs or symptoms suggestive of active TB, no recent close contacts with a person with active TB, and negative QuantiFERON-TB test at screening (if QuantiFERON-TB test is positive, the patient can only be included if active TB is ruled out with appropriate measurements according to standard of care).
* No participation in other clinical trials 4 weeks before and after participation in this study

Exclusion Criteria:

* Concurrent/ongoing treatment with Anakinra (Kineret®) or recent treatment within 3 days prior to screening
* Concurrent/ongoing treatment with other biologics or recent treatment (less than 5 half lives)
* Concurrent/ongoing treatment with

  * oral corticosteroids greater than 10 mg/d within 2 weeks prior to screening
  * parenteral corticosteroids within 4 weeks prior to screening
  * cyclosporin A, methotrexate, dapsone, chloroquine, hydroxychloroquine, azathioprine, cyclophosphamide within 4 weeks prior to screening
  * other immunosuppressives within 4 weeks or 5 half lives prior to screening, whichever is longer
* Evidence of recurrent or latent systemic infection such as tuberculosis
* Significant medical condition rendering the patient immunocompromised or not suitable for a clinical trial
* Treatment with a live (attenuated) virus vaccine during three months prior to Baseline visit (Visit 2)
* An abnormal chest radiograph consistent with clinical signs of prior or present tuberculosis infection whether or not previously treated with anti-tuberculosis agents
* A history of listeriosis, active tuberculosis, persistent chronic or active infection(s) requiring treatment with parenteral antibiotics, parenteral antivirals, or parenteral antifungals within four weeks prior to screening
* Significant concomitant illness such as, but not limited to, cardiac, renal, neurological, endocrinological, metabolic, or lymphatic disease that would adversely affect the subject's participation or evaluation in this study
* Active systemic inflammatory condition other than UV including, but not limited to, rheumatoid arthritis, systemic lupus erythematosus or Sjögren's Syndrome
* History of fibromyalgia or chronic fatigue syndrome
* Evidence of current HIV, active hepatitis B, or hepatitis C infection by clinical or serological history
* History of malignancies within five years prior to screening other than a successfully treated non-metastatic cutaneous, basal, or squamous cell carcinoma and/or in situ cervical cancer
* History of a demyelinating disease or multiple sclerosis
* Severe respiratory disease, including, but not limited to severe bronchiectasis, chronic obstructive pulmonary disease, bullous lung disease, uncontrolled asthma, or pulmonary fibrosis
* Presence of any of the following laboratory abnormalities at enrollment visit: creatinine >1.5 x Upper Limit of Normal (ULN), WBC <3000/µl; platelet count <100000/µl ; ALT or AST >3.0 x ULN
* Lactating females or pregnant females
* Males not willing to use highly effective contraception
* Enrollment in another investigational treatment or device study or use of an investigational agent, or less than 4 weeks or 5 half-lives, whichever is longer, since end of another investigational device or drug trial
* Subjects for whom there is concern about compliance with the protocol procedures
* Any medical condition which, in the opinion of the Investigator, would interfere with participation in the study or place the subject at risk
* History of substance abuse (drug or alcohol) or any other factor (e.g., serious psychiatric condition) that could limit the subject's ability to comply with study procedures
* Subjects who are detained officially or legally to an official institute

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Effect of single doses of canakinumab on the clinical signs and symptoms of urticarial vasculitis measured by the urticarial vasculitis activity score (UVAS) | 18 weeks
  Change in the mean UV activity score (UVAS) from the baseline phase (day -14 to day 0) to the last 2 weeks of the first 4 weeks treatment phase (day 15 to 28) of the study (The UVAS combines the key symptoms of UV). Daily UVAS values will be documented using DHAFs (Daily Health Assessment Forms). Values for the Sum UVAS can range from 0 to 50 per day (5 symptoms, 0-10 each). Mean Daily UVAS will be calculated by dividing the sum of the daily activity scores by 5.

SECONDARY OUTCOMES:
Safety and tolerability following administration of canakinumab to patients with active urticarial vasculitis | 18 weeks
  Safety and tolerability: This includes physical examination, electrocardiogram, routine safety laboratory assessments, clinical observation, vital signs and adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Maurer, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité-Universitätsmedizin Berlin, Berlin, State of Berlin, Germany